CLINICAL TRIAL: NCT05336474
Title: Evaluation of Anatomical and Ultrasonographic Parameters to Predict Difficult Airway in Pediatric Patients
Brief Title: Anatomical and Ultrasonographic Parameters to Predict Difficult Airway in Pediatrics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Demet Altun, Ass. prof., Istanbul University
Other Study IDs: 2020/132
Record Dates: First submitted 2022-04-11; First posted 2022-04-20 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Difficult Airway
Keywords: difficult airway; pediatric anesthesia; laryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonographic upper airway measurements — Ultrasonographic upper airway measurements: Epiglottis-skin distance, Hyoid bone-skin distance, Anterior commissure-skin distance and Thickness of tounge

SUMMARY:
This study was designed to assess the accuracy of ultrasonographic parameters in combination to clinical parameters in the prediction of difficult airway in pediatric population.

All patients underwent a standard airway examination and sonographic airway assessment preoperatively and the predictive values for difficult airway of these methods were recorded.

DETAILED DESCRIPTION:
Difficult airway in a pediatric patient is associated with more stresful situation than adults. Therefore, various clinical airways parameters have been investigated in the prediction of difficult airway. Sonographic evaluation to predict difficult airway is still primitive especially in pediatrics.

Ultrasonography and clinical parameters have been shown to be used in predicting difficult airway, but there is no study showing which is a better predictor.

ELIGIBILITY:
Inclusion Criteria:

* Children, aged between 1-12 years
* Children who required endotracheal intubation under general anesthesia for elective procedures
* written informed parental consent

Exclusion Criteria:

* children over the age of 12
* restrictive neck movement
* tracheostomized patient
* previous laryngeal surgery leading deformation of the laryngeal anatomy

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The patients, aged between 1-12 years, who required endotracheal intubation under general anesthesia for elective procedures were included in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Cormack-Lehane Classification | Three minutes after induction of anesthesia.
  he anesthesiologist, who is blind to the patient's preoperative airway evaluation and ultrasonographic airway measurements, performs intubation and evaluates the laryngeal view.
Epiglottis skin distance in centimeters. | Five minutes before induction of anesthesia.
  The anesthesiologist, who is blind to the patient's preoperative airway evaluation and is experienced user of ultrasonography, measures hyoid bone to skin distance.
Hyoid bone-skin distance in centimeters. | Five minutes before induction of anesthesia.
  The anesthesiologist, who is blind to the patient's preoperative airway evaluation and is experienced user of ultrasonography, measures hyoid bone to skin distance.
Anterior commissure-skin distance in centimeters. | Five minutes before induction of anesthesia
  The anesthesiologist, who is blind to the patient's preoperative airway evaluation and is experienced user of ultrasonography, measures anterior commissure to skin distance.
Thickness of tongue root in centimeters | Five minutes before induction of anesthesia
  The anesthesiologist, who is blind to the patient's preoperative airway evaluation and is experienced user of ultrasonography, measures thickness of tongue root.

SECONDARY OUTCOMES:
intubation difficulty score (IDS )(between 0 to 7) | During the intubation period
  The anesthesiologist, who performed the intubation, evaluated the intubation difficulty.
Mallampati classification | The day before surgery
  Evaluated by the anesthesiologist who performs intubation.
Neck circumference in centimeters. | The day before surgery
  Evaluated by the anesthesiologist who performs intubation.
Sternomental distance in centimeters. | The day before surgery
  The distance between sternal notch and mentum. Evaluated by the anesthesiologist who performs intubation.
Thyromental distance in centimeters | The day before surgery
  The distance between thyroid notch and mentum. Evaluated by the anesthesiologist who performs intubation.
Body mass index (BMI) | The day before surgery
  Weight and height will be combined to report BMI in kg/m^2.Evaluated by the anesthesiologist who performs intubation.
intubation techniques | During the intubation period
  techniques consisting of classic laryngoscope, videolaryngoscope, stylet, and supraglottic airway device used in intubation

CONTACTS AND LOCATIONS:
Overall Officials: Demet Altun, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Inal MT, Memis D, Sahin SH, Gunday I. [Comparison of different tests to determine difficult intubation in pediatric patients]. Rev Bras Anestesiol. 2014 Nov-Dec;64(6):391-4. doi: 10.1016/j.bjan.2014.02.001. Epub 2014 Aug 28. Portuguese. PMID 25437694